CLINICAL TRIAL: NCT07092228
Title: Evaluation of Exercise Capacity in Teenage Females With Abdominal Obesity Using Virtual Reality and Plyometric Workout: Randomized Clinical Trial
Brief Title: Evaluation of Exercise Capacity in Teenage Females Using Virtual Reality and Plyometric Workout
Acronym: VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Ismailia National University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Moeim Abo EL Ros, Assistant Professor of Pediatric Physical Therapy, New Ismailia National University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 3/6/2024- 2025
Record Dates: First submitted 2025-06-24; First posted 2025-07-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Obesity
Keywords: virtual reality; plyometric exercises; abdominal obesity; exercise capacity
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant
Masking Description: using computer software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality and plyometrics (Experimental): using immersed virtual reality combined with plyometric exercises for the lower extremity, in addition to abdominal exercises
  Interventions: Device: virtual reality and plyometric workout
- Treadmill and plyometric (Experimental): using a treadmill aerobic training combined with plyometric exercises for the lower extremity, in addition to abdominal exercises
  Interventions: Device: virtual reality and plyometric workout

INTERVENTIONS:
Device: virtual reality and plyometric workout — to evaluate exercise capacity in teenage females with abdominal obesity using virtual reality and plyometric workouts
  Other Names: treadmill aerobic training and plyometric workout

SUMMARY:
to evaluate the efficacy of virtual reality combined with plyometric workout on abdominal obesity in adolescent females

DETAILED DESCRIPTION:
A total sample size of 100 adolescent females will be assigned to the study and will be divided randomly into two study groups, Study Group A and Study Group B, with 50 subjects in each group. Before the start of the protocol (first session) specific parameters will be taken from all assigned adolescent females in the two groups like waist circumference, waist-hip ratio, Body Mass Index, and some pulmonary function tests in the form of inspiratory reserve volume, Expiratory reserve volume, tidal volume, Inspiratory capacity, and vital capacity. Then, study group A underwent an immersive virtual reality technique in addition to plyometric exercise. Study group B was assigned to a treadmill aerobic workout for 10 minutes in addition to plyometric exercises. All mentioned parameters will be measured again after three months of the treatment program

ELIGIBILITY:
Inclusion Criteria:

* Body mass index more than or equal to 30 Kg/cm2
* waist circumference more than 80 cm
* medical history of polycystic ovarian syndrome
* Age from 13 to 18 years

Exclusion Criteria:

* uncontrolled hypertension
* Rheumatoid arthritis
* Any respiratory diseases like Asthma and respiratory infections
* Osteoprosis

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — not required
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
waist circumference in centimeter | 12 weeks
  An objective outcome measure, measured by a tap measurement before and after treatment protocol
waist-hip ratio in centimeter | 12 weeks
  objective measure objective outcome measure, measured by a tap measurement before and after treatment protocol
Body mass index (BMI) in kg/m² | 12 weeks
  objective outcome measure, s calculated by dividing an individual's weight in kilograms by the square of their height in meters. For children and adolescents, BMI values are categorized to assess weight status (underweight, healthy weight, overweight, obese
pulmonary function tests by using electronic spirometry | 12 weeks
  An objective outcome measure like Forced Expiratory Volume in one second. It's a key measurement in spirometry tests, helping to assess lung function and diagnose conditions like asthma

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No